CLINICAL TRIAL: NCT04970472
Title: Bio Clinical Collection of Urothelial Carcinoma
Acronym: MicroBlad
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0070
Record Dates: First submitted 2021-07-08; First posted 2021-07-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Urothelial Carcinoma; Bladder Cancer
Keywords: Urothelial Carcinoma; neoplasm; bladder cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Neoplasms | interventions — Defecation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, stool, blood and saliva samples will be stored. Tumor samples, collected for primary cares using a punch knife, or a small surgery, will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with Urothelial bladder carcinoma: collection of blood, urines, stool and tumor samples
  Interventions: Biological: collection of blood, urines, stool and tumor samples

INTERVENTIONS:
Biological: collection of blood, urines, stool and tumor samples — blood, urines, stool will be collected during routine cares. Tumor samples from surgery will also be stored.

SUMMARY:
The goal of this study is to collect tumor samples, urines, stool and blood from patients with urothelial carcinoma. These samples will be stored in a secure and confidential laboratory of the Toulouse University Hospital.

DETAILED DESCRIPTION:
Recent studies have shown that the bladder also harbors friendly bacteria that are collectively called the microbiome. While the effect of the bladder microbiome to health remains to be more clearly understood, an imbalance in the microbiome is associated with several urinary diseases including overactive bladder and bladder cancer. But whether the microbiome affects the outcome of Bacille Calmette et Guérin (BCG)-immunotherapy or chemotherapy in bladder cancer is still not known.

Researchers at Toulouse University Hospital want to learn as much as possible about bladder cancer. One way to do so is by studying what is in your urines, blood, stool, saliva and in your tumor.

Patients, who will be agree to take part in this study, will have at least about one tablespoon of blood (as a residual of current biological analysis), 1 container of urines, stool and saliva collected before bladder resection.

After transurethral bladder resection or radical cystectomy scheduled as part of the standard of care, some tumor samples might be collected either as fresh tissue or as paraffin embedded tissue and store in a secure and confidential laboratory at Toulouse University Hospital.

The patient's follow up will be schedule as the standard of care and no additional visit will be required for the study. Oncological outcome of each patient will be recorded up to 5 years This is an investigational study in which up to 500 patients will take part in the collection. All patients will be all enrolled at Toulouse University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old
* Patient with suspected or diagnosed Urothelial carcinoma
* Patients who are willing to consent for this protocol.

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Patients under 18 years old
* Patients under guardianship or curators
* Patients unable to sign a free and informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be all enrolled at Toulouse University Hospital during primary cares.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-07-14 (Estimated); Study Completion 2031-07-14 (Estimated)

PRIMARY OUTCOMES:
Collection and long-term collection of blood, urines, stool and tumor samples from patients with Urothelial bladder carcinoma for future biological and/or surrogate marker studies. | Day 0
  Transcriptomic analysis
Collection and long-term collection of blood, urines, stool and tumor samples from patients with Urothelial bladder carcinoma for future biological and/or surrogate marker studies. | during the intervention/procedure/surgery
  Transcriptomic, proteomic and epigenetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Roumiguie, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Rangueil University Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No